CLINICAL TRIAL: NCT06521034
Title: Omprehensive First-in-Human Phase I/II Study of FHND-9041 in Patients With EGFR Mutated Advanced Non-Small Cell Lung Cancer
Brief Title: First-in-Human Phase I/II Study of FHND-9041 in Patients With EGFR Mutated Advanced Non-Small Cell Lung Cancer
Acronym: Helpful
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yongchang Zhang (Other)
Collaborators: Jiangsu Chia Tai Fenghai Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yongchang Zhang, Professor, Director of Clinical Trial Center, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018L0290
Record Dates: First submitted 2024-07-15; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer; EGFR Gene Mutation; EGFR-TKI Sensitizing Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (arm A, Dose Escalation Study) (Experimental): In Phase I, patients with NSCLC harboring the EGFRT790M mutation and prior failure with EGFR-TKIs were enrolled. Using a "3+3" design, dose escalation and expansion studies were conducted to evaluate the safety and pharmacokinetics of FHND-9041 at doses of 40, 80, 120, and 180 mg/day, with 3 to 9 patients per group. Phase II utilized the RP2D of 80 mg QD, determined from Phase I, to assess the efficacy and safety of FHND-9041 in patients with locally advanced or metastatic NSCLC. The primary endpoint was Objective Response Rate (ORR), with Progression-Free Survival (PFS) as a secondary endpoint. Tumor response and disease progression were evaluated according to RECIST 1.1 criteria, and safety was assessed per CTCAE-5.0 standards.
  Interventions: Drug: FHND-9041
- Treatment Group (arm B, Dose Expansion Study) (Experimental): In Phase Ⅱ, after comprehensive analysis and consultation, at least 30 patients were enrolled according to the inclusion and exclusion criteria. 37 patients with locally advanced or metastatic EGFR-mutated NSCLC receiving first-line treatment were enrolled. Tumor response and disease progression were evaluated according to RECIST 1.1 criteria, and safety was assessed per CTCAE-5.0 standards.
  Interventions: Drug: FHND-9041

INTERVENTIONS:
Drug: FHND-9041 — In Phase I, using a "3+3" design, dose escalation and expansion studies were conducted at doses of 40, 80, 120 and 180 mg/day. At least 3 patients were enrolled in each dose arm, and no dose-limiting toxicities were observed. With a plateau observed at 120 mg/day, the 80 mg/d and 120mg/d groups were selected for dose expansion. The 80mg/d queue has expanded by 36 patients, and the 120mg/d queue has expanded by 39 patients. In Phase Ⅱ, after comprehensive analysis and consultation, at least 30 patients were enrolled according to the inclusion and exclusion criteria. 37 patients with locally advanced or metastatic EGFR-mutated NSCLC receiving first-line treatment were enrolled.
  Other Names: EGFR-TKI

SUMMARY:
FHND-9041 capsule is a novel third-generation EGFR inhibitor targeting EGFR-sensitive mutations. This first-in-human study is a single-arm, multi-center, open-label, non-randomized Phase Ⅰ/II trial. It aims to evaluate the tolerability, safety, pharmacokinetics, and anti-tumor activity of FHND-9041 in patients with NSCLC harboring the EGFRT790M mutation, particularly those acquiring resistance to prior EGFR-TKI treatment. Additionally, the study seeks to determine the Recommended Phase II Dose (RP2D) of FHND-9041and assess its efficacy as a first-line treatment for patients with locally advanced or metastatic NSCLC harboring EGFR-sensitive mutations.

DETAILED DESCRIPTION:
FHND-9041 capsule is a novel third-generation EGFR inhibitor targeting EGFR-sensitive mutations. This first-in-human study is a single-arm, multi-center, open-label, non-randomized Phase Ⅰ/II trial. It aims to evaluate the tolerability, safety, pharmacokinetics, and anti-tumor activity of FHND-9041 in patients with NSCLC harboring the EGFRT790M mutation, particularly those acquiring resistance to prior EGFR-TKI treatment. Additionally, the study seeks to determine the Recommended Phase II Dose (RP2D) of FHND-9041and assess its efficacy as a first-line treatment for patients with locally advanced or metastatic NSCLC harboring EGFR-sensitive mutations. The primary end point was Pharmacokinetic Parameters and secondary endpoints was ORR and PFS etc.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria for study eligibility:

  1. Subjects who have fully understood the trial and are willing to sign the informed consent form.
  2. Age of at least 18 years and not more than 75, with no gender restrictions.
  3. NSCLC diagnosed by histology or cytology.
  4. Patients diagnosed with locally advanced or metastatic NSCLC who are not suitable for surgery or radiotherapy.
  5. Previous treatment and mutation types:

  <!-- -->

  1. Subjects enrolled in the group of the second or third-line treatment patients with EGFR T790M mutations should have previously existed sensitive mutations (including Del l9, L858R, etc) and have previously received an EGFR-TKI (such as gefitinib, erlotinib, icotinib or afatinib) and experienced disease progression, and a written test report should confirm the occurrence of EGFR T790M mutation.
  2. Subjects enrolled in the group of the first-line treatment patients with EGFRm+ should have not received systemic treatment regimen, including chemotherapy and/or EGFR-TKI, and a written test report should confirm the detection of EGFR sensitive mutations (including exon 19 deletion or L858R, both alone or co-existing with other EGFR site mutations). Patients who had received previous adjuvant or neoadjuvant therapy (chemotherapy, radiotherapy, or other treatment) were eligible if they had not progressed one year after the end of treatment and patients who had received local therapy (radiotherapy or pleural perfusion) were eligible to participate if the lesions within the scope of local therapy were nontarget 6. Baseline at least one tumor lesions can meet the following requirements: (1) always without radiation exposure, also not used to screen period biopsy (if only one measurable lesion, participants can accept needle aspiration cytology and biopsy examination genetic status confirmation, but as a baseline imaging studies should be carried out in puncture inspection at least 7 days). (2) The maximum diameter of the baseline stage should be ≥10mm (if it is lymph node, the short axis should be ≥15mm); (3) CT or MRI, but need to use the same method at follow-up evaluation。 7. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2 and an expected survival time of at least 3 months.

  8. Subjects have at least one measurable lesion that meets the RECIST version 1.1 criteria.

  9. If female subjects of childbearing potential, they must take adequate contraception measures (such as condoms) throughout the trial and for 3 months after the last administration of the trial drug. A negative pregnancy test should be obtained prior to drug administration.

  10. Male subjects must agree to use barrier contraceptive measures (such as condoms) during the test period for 6 months after the last administration of the trial drug.

  11. Patients were able to agree and proceed with planned visits, treatments, laboratory tests, and other study procedures.

Exclusion Criteria:

-

The following conditions make subjects ineligible to participate in this study:

1. Patients had received any cytotoxic chemotherapy in a previous regimen or clinical study within 14 days before the first dose and patients who had not previously received any EGFR-TKI were required to be enrolled in the EGFRm+ first-line treatment group.
2. The interval between the last treatment with EGFR-TKI (such as erlotinib, gefitinib, afatinib, or osimertinib) and the first administration of the study drug is less than 5 half-lives, and the specific drug involved is determined by the researcher's comprehensive consideration.
3. The interval between the last treatment with other experimental drugs or anticancer drugs and the first administration of the study drug is less than 5 half-lives
4. The patient had used the third generation EGFR-TKI drugs (such as AZD9291, CO-1686, HM61713, ASP8273, EGF816, mevalatinib, ivirinib, eflutinib, etc.) or their raw materials or generic drugs
5. A confirmed EGFR exon 20 insertion mutation was present at any time after the initial diagnosis.
6. The subject has undergone major surgery (including vascular access establishment); patients who received radiation to more than 30% of the bone marrow or large field radiation within 4 weeks before the first administration of the study treatment.
7. Subjects who are currently using or have used drugs or herbal supplements known to be strong inhibitors or inducers of CYP3A4 and CYP2C8 within 1 week (Appendix 3).
8. At the start of the study treatment, toxic reactions from previous treatment are still present and exceed grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE), except for hair loss. The previous platinum treatment-related neurotoxicity may be relaxed to grade 2.
9. Patients with symptomatic spinal cord compression or brain metastasis, stable disease without symptoms, and who do not require corticosteroid treatment within 4 weeks before the start of the study treatment, except for those who require treatment for the above conditions.
10. Any clinical evidence suggesting severe or uncontrolled systemic diseases, such as patients who are not suitable for participation in the trial as judged by the investigator or who have uncontrolled hypertension and active bleeding tendencies that may affect compliance with this clinical trial, as well as active infections, such as hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection.
11. The average corrected QT interval (QTc) obtained from 3 electrocardiogram (ECG) examinations in a resting state is >470 msec (the first ECG indicates abnormal, and 2 repeat measurements are taken to obtain the average corrected value).
12. Various severe and clinically significant abnormalities in heart rhythm, conduction, and resting ECG morphology, such as complete left bundle branch block, third-degree atrioventricular block, second-degree atrioventricular block, PR interval >250 msec, and so on.
13. Various factors that may increase the risk of QTc prolongation or arrhythmia events, such as heart failure, hypokalemia (except for those who have been treated with potassium supplementation and re-examined normally before the first administration), congenital long QT syndrome, a family history of long QT syndrome or unexplained sudden death before the age of 40, and various combined medications that may prolong the QT interval.
14. A history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid treatment, or active interstitial lung disease clinically.
15. Bone marrow reserve or organ dysfunction with the following laboratory values: absolute neutrophil count <1.5×10^9/L; platelet count <100×10^9/L; hemoglobin <90g/L; if there is no clear evidence of liver metastasis, aspartate aminotransferase (ALT) >2.5 times the upper limit of normal (ULN); if there is liver metastasis, ALT>5 times ULN; if there is no clear evidence of liver metastasis, alanine aminotransferase (AST) >2.5 times ULN; if there is liver metastasis, AST>5 times ULN; if there is no liver metastasis, total bilirubin >1.5 times ULN; if there is Gilbert syndrome (unconjugated hyperbilirubinemia) or liver metastasis, total bilirubin >3 times ULN; or creatinine greater than 1.5 × ULN concurrent with creatinine clearance less than 50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance was required only when creatinine was greater than 1.5 × ULN.
16. The drug can't stability control of high blood sugar.
17. Patients who received blood transfusion within 2 weeks before screening;
18. Uncontrollable nausea and vomiting, chronic gastrointestinal diseases, and patients who cannot swallow drug preparations, and have undergone extensive intestinal resection surgery may affect the full absorption of FHND-9041.
19. Subjects with a history of hypersensitivity reactions to the excipients of FHND-9041.
20. There are other patients with malignant tumor or other malignant tumor diagnosis in recent five years before (except basal cell carcinoma or cervical breast carcinoma in situ).
21. Female subjects who are breastfeeding.
22. According to the researchers' judgment, if the subject cannot comply with the study procedures, regulations, and requirements, they cannot participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters of Maximum Serum Concentration (Cmax) after cycle 1 | through study completion, an average of 1 year
  Maximum serum concentration (Cmax) in patients with locally advanced or metastatic EGFR T790M mutation non-small cell lung cancer (NSCLC) who treated with FHND-9041.
Pharmacokinetic Parameters Area Under the Concentration-Time Curve After Cycle 1 | through study completion, an average of 1 year
  Area under the concentration versus-time curve from time 0 to the last quantifiable concentration (AUClast) and during the dosing interval (AUCtau) of FHND-9041 was assessed.

SECONDARY OUTCOMES:
Objective Response Rate | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 12 months post-dose
  Objective response rate (ORR) was defined as unconfirmed complete response (CR) and partial response (PR) as assessed by the investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Treatment-Emergent Adverse Events of Any Grade by System Organ Classes | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to approximately 12 months post-dose
  Adverse events (AEs) were to be coded using MedDRA Version 20.1 and assigned severity grades based on Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. A treatment-emergent adverse event (TEAE) was defined as an AE that occurred, having been absent before the first dose of study drug, or had worsened in severity or seriousness after initiating the study drug after last dose of study drug.
Progression free survival | Time from first subject dose to study completion, or up to 36 month
  Progression-free survival (PFS) is defined as the time from random assignment to disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No